CLINICAL TRIAL: NCT01488201
Title: A Randomized, Placebo-controlled, Ascending Single-dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of KHK4827 in Healthy Volunteers and Subjects With Moderate to Severe Psoriasis
Brief Title: A Clinical Pharmacology of KHK4827 in Healthy Volunteers and Subject With Moderate to Severe Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4827-001
Record Dates: First submitted 2011-12-01; First posted 2011-12-08 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2012-11

CONDITIONS: Psoriasis
Keywords: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — brodalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- KHK4827 (Experimental)
  Interventions: Drug: KHK4827
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: KHK4827
  Arms: KHK4827

SUMMARY:
This is a randomized, placebo-controlled, ascending single dose study of KHK4827 to evaluate safety, tolerability, pharmacokinetics and pharmacodynamics of subcutaneous or intravenous administration of KHK4827 in healthy male subjects or moderate to severe psoriasis patients.

ELIGIBILITY:
Inclusion Criteria:

Health volunteers

* Able to provide written informed consent
* Healthy male between 20 to 45 years of age, inclusive at the time of screening
* Additional inclusion criteria apply

Psoriasis subjects

* 20 to 70 years of age, inclusive at the time of screening
* Active but clinically stable, plaque psoriasis
* Psoriasis involving ≥10% of the body surface area
* A minimum PASI score of ≥10 obtained during the screening period
* Additional inclusion criteria apply

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Safety
  * Adverse events
  * Clinical laboratory test data
  * Vital signs

SECONDARY OUTCOMES:
Plasma KHK4827 concentrations and pharmacokinetic parameters | 16 time points up to 64 days
  To assess PK parameters which include
  * area under the plasma concentration versus time curve (AUC)
  * peak plasma concentration (Cmax)
  * t1/2
  * CL

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo, Japan